CLINICAL TRIAL: NCT02967068
Title: VCRC Tissue Biorepository Collection Protocol
Brief Title: VCRC Tissue Repository
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Office of Rare Diseases (ORD) (NIH)
Responsible Party: Principal Investigator, Peter Merkel, Chief, Division of Rheumatology Professor of Medicine and Epidemiology, University of Pennsylvania
Other Study IDs: VCRC5511; U54AR057319 (NIH)
Record Dates: First submitted 2016-11-11; First posted 2016-11-17 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Aortitis; Cutaneous Vasculitis; Eosinophilic Granulomatosis With Polyangiitis; Giant Cell Arteritis; Granulomatosis With Polyangiitis (Wegener's); Henoch-Schonlein Purpura; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis; Churg-Strauss Syndrome
Keywords: CSS; EGPA; GCA; GPA; MPA; PAN; TAK; HSP
MeSH Terms: conditions — Aortitis; Skin Diseases, Vascular; Churg-Strauss Syndrome; Giant Cell Arteritis; Granulomatosis with Polyangiitis; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biopsy specimens collected as standard of care for these diseases will be retrieved and used in research. The most common biopsies performed are kidney, lung, skin, nerves, and vessels.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to collect existing tissue specimens from subjects enrolled in Vasculitis Clinical Research Consortium (VCRC) studies. Analysis of these tissue specimens and linked clinical data collected through VCRC studies may lead to the identification and development of a series of translational research projects. Results of these studies will provide vasculitis researchers with insight into the causes of these diseases and generate new ideas for diagnostic tests and therapies, and will be of great interest to the larger communities of researchers investigating vasculitis and other autoimmune, inflammatory, and vascular diseases.

DETAILED DESCRIPTION:
Biopsy specimens collected as standard of care for these diseases will be retrieved and used in research. The most common biopsies performed are kidney, lung, skin, nerves, and vessels; however, other tissue is also of interest for the study. Biopsies are not performed as part of this protocol, rather we will request consent to collect biopsy specimens already collected under routine care.

ELIGIBILITY:
Inclusion Criteria:

* A participant will be deemed eligible for this study if the participant is/was enrolled in another one of the VCRC observational/longitudinal protocols (5502, 5503, 5504, 5505, 5506, 5507, 5563) and/or one of the VCRC interventional studies (5522, 5523, 5526, 5527, or 5562).

Exclusion Criteria:

* Inability to give informed consent (or their guardians in the case of children) and to sign the consent form.
* Unwilling to allow the use of their tissue for research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1000 patients with GCA, TAK, PAN, GPA, MPA, EGPA, cutaneous vasculitis and aortitis will potentially be enrolled into the VCRC Tissue Biorepository Collection Protocol.
  The protocol will be conducted at the major vasculitis centers in the United States and Canada participating in selected VCRC studies. Biopsy specimens collected as standard of care for these diseases will be retrieved and used in research.
  Biopsies are not performed as part of this protocol, rather we will request consent to collect biopsy specimens already collected under routine care.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Identify genes that increase the risk of developing vasculitis | 1 year
  Evaluating of clinical data and linked biopsy specimens to identify genes that increase the risk of developing vasculitis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (8):
- United States (6):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - University of Toronto Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/vcrc/
- See also: Rare Diseases Clinical Research Network — http://rarediseasesnetwork.org